CLINICAL TRIAL: NCT01867333
Title: A Randomized Phase II Trial Combining Vaccine Therapy With PROSTVAC /TRICOM and Enzalutamide vs. Enzalutamide Alone in Men With Metastatic Castration Resistant Prostate Cancer
Brief Title: Enzalutamide With or Without Vaccine Therapy for Advanced Prostate Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Ravi A. Madan, M.D., Principal Investigator, National Cancer Institute (NCI)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 130146; 13-C-0146
Record Dates: First submitted 2013-05-30; First posted 2013-06-04 (Estimated); Results first posted 2023-09-26 (Actual); Last update posted 2023-09-26 (Actual); Status verified 2023-09

CONDITIONS: Prostate Cancer
Keywords: Immunotherapy; Gene Transfer; Androgen Receptor Antagonist; PSA; Immune Response
MeSH Terms: conditions — Prostatic Neoplasms | interventions — PROSTVAC; enzalutamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm 1 - Enzalutamide alone (Experimental): Enzalutamide alone. Enzalutamide will be given at the standard dose of 160 mg daily.
  Interventions: Biological: Enzalutamide
- Arm 2 - Enzalutamide with Prostate-Specific Antigen (PSA)-TRICOM (Experimental): Enzalutamide with PSA-TRICOM. Enzalutamide will be given at the standard dose of 160 mg daily with vaccine given week 1 (vaccinia-PSA-TRICOM, 2x10(8) infectious units subcutaneously) and then week 3, 5 and then monthly fowlpox-vaccine (1x10(9) infectious units subcutaneously).
  Interventions: Biological: PROSTVAC (rilimogene galvacirepvec/rilimogene glafolivec) -F/TRICOM; Biological: PROSTVAC (rilimogene galvacirepvec/rilimogene glafolivec) -V/TRICOM; Biological: Enzalutamide

INTERVENTIONS:
Biological: PROSTVAC (rilimogene galvacirepvec/rilimogene glafolivec) -F/TRICOM — A recombinant fowlpox virus vector vaccine containing the genes for human prostate-specific antigen (PSA) and three co-stimulatory molecules.
  Arms: Arm 2 - Enzalutamide with Prostate-Specific Antigen (PSA)-TRICOM
Biological: PROSTVAC (rilimogene galvacirepvec/rilimogene glafolivec) -V/TRICOM — A recombinant vaccinia virus vector vaccine containing the genes for human prostate-specific antigen (PSA) and three co-stimulatory molecules.
  Arms: Arm 2 - Enzalutamide with Prostate-Specific Antigen (PSA)-TRICOM
Biological: Enzalutamide — An androgen receptor inhibitor.
  Other Names: Xtandi

SUMMARY:
Background:

- Enzalutamide is a hormone therapy that is used to treat advanced prostate cancer. It is given after chemotherapy and surgery to help the body destroy the cancer cells. A new possible way of treating prostate cancer is using a vaccine that may help stimulate the immune system. It will help white blood cells recognize and kill the cancer cells in and around the prostate. Researchers want to see whether this vaccine, given with enzalutamide, is more effective at treating advanced prostate cancer than enzalutamide alone.

Objectives:

- To compare the safety and effectiveness of enzalutamide with and without vaccine therapy for advanced prostate cancer.

Eligibility:

- Men at least 18 years of age who have advanced castration-resistant prostate cancer.

Design:

* Participants will be screened with a physical exam and medical history. Blood and urine samples will be collected. Imaging studies will be used to monitor the cancer before treatment.
* Participants will be separated into two groups. One group will have enzalutamide and the study vaccine. The other group will have enzalutamide alone.
* All participants will take enzalutamide once a day. They will take the drug during 4-week cycles of treatment.
* Treatment will be monitored with frequent blood tests and imaging studies. Participants will continue to take the study drug for as long as the cancer does not grow, and the side effects are not severe.
* The vaccine group of participants will also have the new study vaccine. They will have a single injection on the first day of the first study cycle. There will be regular booster injections afterward. There will be one on day 15 of the first cycle, the first day of the second cycle. The vaccine will then be given every 4 weeks for the next four cycles, and then every 12 weeks (every 3 cycles) thereafter. Participants will continue to have the study vaccine for as long as the cancer does not grow, and the side effects are not severe.

DETAILED DESCRIPTION:
Background:

* Enzalutamide is a well-tolerated, modern androgen receptor antagonist (ARA) with more enhanced anti-tumor activity compared to previous ARAs. Phase III trial has demonstrated a 4.8 month improvement in survival and a 37% risk reduction in death in metastatic castration resistant prostate cancer (mCRPC) patients who have had previous docetaxel.
* PROSTVAC is a therapeutic cancer vaccine which is designed to induce an anti-tumor immune response. In a randomized controlled Phase 2 trial, PROSTVAC (rilimogene galvacirepvec/rilimogene glafolivec) therapy was associated with a prolongation of survival by 8.5 months in men with metastatic castrate-resistant prostate cancer. An international Phase 3 trial is on-going.
* Preclinical data has demonstrated that hormonal therapies such as ARAs can enhance the immune response through multiple mechanisms. Specifically, our group has shown that enzalutamide can increase thymic production of na(SqrRoot) ve T-cells, which could be activated by a cancer vaccine. Together, these data provide an important rationale to combine enzalutamide with PSA-TRICOM in mCRPC.
* Data from the clinical trials with these therapies suggest that they are very well tolerated and without overlapping toxicity.

Objective:

-Determine if prostate-specific antigen (PSA)-TRICOM combined with enzalutamide will increase time to progression (as defined by Prostate Cancer Clinical Trials Working Group 2 criteria, incorporated in section 5.2) in chemotherapy-naive metastatic castration resistant prostate cancer patients compared to enzalutamide alone.

Design:

* The study will randomize chemotherapy-naive, mCRPC patients to either enzalutamide alone or enzalutamide with PSA-TRICOM. Enzalutamide will be given at the standard dose of 160 mg daily.
* PSA-TRICOM will be administered identical to the Phase III dosing with vaccine given week 1 (vaccinia-PSA-TRICOM, 2x10(8) units subcutaneously) and then week 3, 5 and then monthly fowlpox-vaccine (1x10(9) units subcutaneously).
* After completing 6 months of vaccine, fowlpox-vaccine (1x10(9) units subcutaneously will be administered every 3 months. Patients will be treated until radiographic progression on scans using Prostate Cancer Working Group Criteria.

Eligibility:

* mCRPC patients with rising PSA or progressive disease despite castration levels of testosterone.
* Chemotherapy-na(SqrRoot) ve with minimal or no symptoms related to prostate cancer.
* Patients with history of autoimmune disease, brain/leptomeningeal metastasis, a second malignancy within 3 years of enrollment, or a severe co-morbid condition will be excluded.
* Patients who have received abiraterone will be excluded
* Patients will be stratified based on previous immunotherapy used as cancer treatment.

ELIGIBILITY:
* INCLUSION CRITERIA:
* Patients must have histologically or cytologically confirmed prostate cancer confirmed by either the Laboratory of Pathology at the National Institutes of Health (NIH) Clinical Center or Walter Reed National Military Medical Center at Bethesda prior to starting this study. If no pathologic specimen is available, patients may enroll with a pathologist's report showing a histological diagnosis of prostate cancer and a clinical course consistent with the disease.
* Castrate testosterone level (<50ng/dl or 1.7nmol /L)
* Metastatic disease documented by one of the following:
* Metastatic bone disease on an imaging study, or
* Soft tissue disease documented by computed tomography (CT)/magnetic resonance imaging (MRI), or
* Progressive disease at study entry defined as one or more of the following criteria occurring in the setting of castrate levels of testosterone:

  i. Radiographic progression defined as any new or enlarging bone lesions or growing lymph node disease, consistent with prostate cancer OR

ii. Prostate-specific antigen (PSA) progression defined by sequence of rising values separated by >1 week (2 separate increasing values over a minimum of 2ng/ml (Prostate Cancer Clinical Trials Working Group (PCWG2) PSA eligibility criteria). If patients had been on flutamide, PSA progression is documented 4 weeks or more after withdrawal.

The requirement for a 4-6 weeks withdrawal period following discontinuation of flutamide, nilutamide or bicalutamide only applies to patients who have been on these drugs for at least the prior 6 months. For all other patients they must stop bicalutamide, nilutamide or flutamide the day prior to enrollment.

* Asymptomatic or mildly symptomatic from prostate cancer; no use of regularly scheduled opiate analgesics for prostate cancer-related pain
* Patients must agree to continue to continuation of androgen deprivation therapy (ADT) with a gonadotropin-releasing hormone analogue/antagonist or bilateral orchiectomy
* Age greater than or equal to 18 years.
* Eastern Cooperative Oncology Group (ECOG) performance status less than or equal to 1 (Karnofsky greater than or equal to 80%).
* Patients must have normal organ and marrow function as defined below:
* absolute neutrophil count greater than or equal to 1,500/mcL
* platelets greater than or equal to 100,000/mcL
* total bilirubin within normal institutional limits; for patients with Gilbert's syndrome, total bilirubin less than or equal to 3.0mg/dL
* Aspartate aminotransferase (AST) serum glutamic-oxaloacetic transaminase (SGOT)/alanine aminotransferase (ALT) serum glutamic pyruvic transferase (SGPT) less than or equal to 2.5 times institutional upper limit of normal
* creatinine within 1.5 X normal institutional limits, OR
* creatinine clearance greater than or equal to 60 mL/min/1.73 m(2) for patients with creatinine levels above institutional normal by Cockcroft-Gault Equation
* The effects of enzalutamide alone or in combination with PSA-TRICOM on the developing human fetus are unknown. For this reason, men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation and for three (3) months after the last dose of enzalutamide. Should a woman become pregnant or suspect she is pregnant while her partner is participating in this study, she should inform her treating physician immediately.
* Ability of subject to understand and the willingness to sign a written informed consent document.

EXCLUSION CRITERIA:

* Patients who are immunocompromised as listed as follows:
* Human immunodeficiency virus positivity due to the potential for decreased tolerance and may be at risk for severe side effects
* Chronic administration (defined as daily or every other day for continued use >14 days) of systemic corticosteroids (including steroid eye drops) or other immune suppressive drugs, within 28 days before the first planned dose of PSA-TRICOM. Nasal, or inhaled steroid, and topical steroid creams for small body areas are not excluded.
* Patients who have undergone allogeneic peripheral stem cell transplantation, or solid organ transplantation requiring immunosuppression
* History of splenectomy
* History of, or active autoimmune disease (such as Autoimmune neutropenia, thrombocytopenia, or hemolytic anemia, systemic lupus erythematosis, Sjogrens syndrome, scleroderma, myasthenia gravis, Goodpasture's syndrome, Addisons disease, Hashimoto's thyroiditis, Crohn's or Grave's disease). Patients with type 1 diabetes mellitus or vitiligo are not excluded if the condition is well controlled.
* Patients with a history of brain/leptomeningeal metastasis
* Patients who have been treated with abiraterone will be excluded
* Patients with history of seizure as an adult including febrile seizure or any condition that may predispose to seizure (e.g., prior stroke, brain arteriovenous malformation, head trauma with loss of consciousness requiring hospitalization). Also, current or prior treatment with anti-epileptic medications for the treatment of seizures or history of loss of consciousness. Also transient ischemic attack within 12 months prior to randomization will not be permitted.
* Patients with second malignancy within 3 years of enrollment; Patients curatively treated non-melanoma skin cancers or carcinoma in situ of the bladder, are not excluded.
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to enzalutamide or poxviral vaccines (e.g., vaccinia vaccine)
* Known allergy to eggs, egg products, aminoglycoside antibiotics (for example, gentamicin or tobramycin),
* History of atopic dermatitis or active skin condition (acute, chronic, exfoliative) that disrupts the epidermis
* Previous adverse reactions to smallpox vaccination
* Unable to avoid close contact or household contact with the following high-risk individuals for three weeks after the Day 1 vaccination: (a) children less than or equal to 3 years of age, (b) pregnant or nursing women, (c) individuals with prior or concurrent extensive eczema or other eczematoid skin disorders, or (d) immunocompromised individuals, such as those with human immunodeficiency virus (HIV).
* Any condition which, in the opinion of the investigator, would prevent full participation in this trial (including the long-term follow-up), or would interfere with the evaluation of the trial endpoints.
* Patients with prior chemotherapy for nonmetastatic prostate cancer within a year are excluded.
* Receipt of an investigational agent within 28 days (or 56 days for an antibody-based therapy) before the first planned dose of study drugs. (Immune checkpoint inhibitors that are antibody-based will only require 28 days before enrollment)
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, uncontrolled hypertension (systolic blood pressure (SBP)>170/ diastolic blood pressure (DBP)>105) or psychiatric illness/social situations within 12 months that would limit compliance with study requirements.
* Use of herbal products that may decrease PSA levels (e.g., saw palmetto)
* Any gastrointestinal disease that could hinder the absorption of enzalutamide.
* Patients who have had chemotherapy for metastatic castration-resistant prostate cancer. (Patients who have had docetaxel for metastatic castration sensitive disease per Chemo-hormonal Therapy versus Androgen Ablation Randomized Trial for Extensive Disease (CHAARTED) Data35 may enroll as long as they did not have progressive disease while on docetaxel and are 6 months removed from treatment, with all treatment related toxicities resolving to at least grade 1.)
* Patients who have received radiation therapy, radionuclide therapy or undergone surgery within certain duration (4 weeks) of enrollment

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2013-08-12 (Actual); Primary Completion 2022-09-28 (Actual); Study Completion 2022-10-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ravi A Madan, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
All individual participant data (IPD) recorded in the medical record will be shared with intramural investigators upon request. In addition, all large-scale genomic sequencing data will be shared with subscribers to the database of Genotypes and Phenotypes (dbGaP).
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Clinical data available during the study and indefinitely. Genomic data are available once genomic data are uploaded per protocol Genomic Data Sharing (GDS) plan for as long as the database is active.
Access Criteria: Clinical data will be made available via subscription to Translational Research Information System (BTRIS) and with permission of the study principal investigator (PI). Genomic data are made available via the database of Genotypes and Phenotypes (dbGaP) through requests to the data custodians

REFERENCES:
- [Background] Kantoff PW, Schuetz TJ, Blumenstein BA, Glode LM, Bilhartz DL, Wyand M, Manson K, Panicali DL, Laus R, Schlom J, Dahut WL, Arlen PM, Gulley JL, Godfrey WR. Overall survival analysis of a phase II randomized controlled trial of a Poxviral-based PSA-targeted immunotherapy in metastatic castration-resistant prostate cancer. J Clin Oncol. 2010 Mar 1;28(7):1099-105. doi: 10.1200/JCO.2009.25.0597. Epub 2010 Jan 25. PMID 20100959
- [Background] Madan RA, Arlen PM, Mohebtash M, Hodge JW, Gulley JL. Prostvac-VF: a vector-based vaccine targeting PSA in prostate cancer. Expert Opin Investig Drugs. 2009 Jul;18(7):1001-11. doi: 10.1517/13543780902997928. PMID 19548854
- [Background] Scher HI, Fizazi K, Saad F, Taplin ME, Sternberg CN, Miller K, de Wit R, Mulders P, Chi KN, Shore ND, Armstrong AJ, Flaig TW, Flechon A, Mainwaring P, Fleming M, Hainsworth JD, Hirmand M, Selby B, Seely L, de Bono JS; AFFIRM Investigators. Increased survival with enzalutamide in prostate cancer after chemotherapy. N Engl J Med. 2012 Sep 27;367(13):1187-97. doi: 10.1056/NEJMoa1207506. Epub 2012 Aug 15. PMID 22894553
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2013-C-0146.html
- See also: http://www.clinicaltrials.gov — http://www.clinicaltrials.gov

RESULTS

PARTICIPANT FLOW:
Groups:
- Arm 1 - Enzalutamide Alone: Enzalutamide alone
  Enzalutamide: An androgen receptor inhibitor.
  Enzalutamide will be given at the standard dose of 160 mg daily.
- Arm 2 - Enzalutamide With Prostate-Specific Antigen (PSA)-TRICOM: Enzalutamide with PSA-TRICOM
  PROSTVAC (rilimogene galvacirepvec/rilimogene glafolivec) -F/TRICOM: A recombinant fowlpox virus vector vaccine containing the genes for human prostate-specific antigen (PSA) and three co-stimulatory molecules.
  PROSTVAC (rilimogene galvacirepvec/rilimogene glafolivec) -V/TRICOM: A recombinant vaccinia virus vector vaccine containing the genes for human prostate-specific antigen (PSA) and three co-stimulatory molecules.
  Enzalutamide: An androgen receptor inhibitor.
  Enzalutamide will be given at the standard dose of 160 mg daily with vaccine given week 1 (vaccinia-PSA-TRICOM, 2x10(8) infectious units subcutaneously) and then week 3, 5 and then monthly fowlpox-vaccine (1x10(9) infectious units subcutaneously).
Period: Overall Study
Arm/Group | Arm 1 - Enzalutamide Alone | Arm 2 - Enzalutamide With Prostate-Specific Antigen (PSA)-TRICOM
Started | 29 | 28
Completed | 21 | 23
Not Completed | 8 | 5
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Adverse Event | 1 | 0
Not completed — Participant choice | 1 | 2
Not completed — Complicating disease/intercurrent illness | 1 | 0
Not completed — Death | 0 | 1
Not completed — Physician Decision | 3 | 2
Not completed — Switched to alternative treatment | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm 1 - Enzalutamide Alone | Arm 2 - Enzalutamide With Prostate-Specific Antigen (PSA)-TRICOM | Total
Number analyzed (Participants) | 29 | 28 | 57
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 11 | 13 | 24
  >=65 years | 18 | 15 | 33
Age, Continuous [Mean (Standard Deviation); unit: years] | 67.78 (10.72) | 67.12 (10.61) | 67.45 (10.58)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 29 | 28 | 57
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1
  Not Hispanic or Latino | 28 | 28 | 56
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 5 | 5 | 10
  White | 22 | 23 | 45
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 29 | 28 | 57

OUTCOME MEASURES:

1. Primary Outcome: Time to Progression (TTP)
Description: Time to progression is defined as the duration of time from start of treatment to time of disease progression. Progression was measured by the Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1. Progression is defined as at least a 20% increase in the sum of the diameters of target lesions, taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study). The appearance of one or more new lesions can also be considered progression if they meet the size criteria for target lesions.
Time Frame: Median follow-up of 55.4 months
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Arm 1 - Enzalutamide Alone | Arm 2 - Enzalutamide With Prostate-Specific Antigen (PSA)-TRICOM
Number analyzed (Participants) | 29 | 28
Months | 24.2 [16.6 to 33.1] | 19.1 [8.5 to 30.3]

2. Secondary Outcome: Overall Survival
Description: Overall survival is defined as the date of on-study to the date of death from any cause or last follow up.
Time Frame: Median potential follow-up of 68.5 months
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Arm 1 - Enzalutamide Alone | Arm 2 - Enzalutamide With Prostate-Specific Antigen (PSA)-TRICOM
Number analyzed (Participants) | 29 | 28
Months | 45.6 [26.9 to 54.7] | 33.8 [20.0 to 73.2]

3. Secondary Outcome: Time to Prostate-specific Antigen (PSA) Progression
Description: PSA progression is defined by a sequence of rising values separated by >1 week (2 separate increasing values over a minimum of 2ng/ml or 25% higher (Prostate Cancer Clinical Trials Working Group (PCWG2) PSA eligibility criteria).
Time Frame: Median follow-up of 55.4 months
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Arm 1 - Enzalutamide Alone | Arm 2 - Enzalutamide With Prostate-Specific Antigen (PSA)-TRICOM
Number analyzed (Participants) | 29 | 28
Months | 11 [6.4 to 17.5] | 16 [4.6 to 38.6]

4. Other Pre Specified Outcome: Number of Participants With Serious and/or Non-serious Adverse Events Assessed by the Common Terminology Criteria for Adverse Events (CTCAE v4.0)
Description: Here is the number of participants with serious and/or non-serious adverse events assessed by the Common Terminology Criteria for Adverse Events (CTCAE v4.0). A non-serious adverse event is any untoward medical occurrence. A serious adverse event is an adverse event or suspected adverse reaction that results in death, a life-threatening adverse drug experience, hospitalization, disruption of the ability to conduct normal life functions, congenital anomaly/birth defect or important medical events that jeopardize the patient or subject and may require medical or surgical intervention to prevent one of the previous outcomes mentioned.
Time Frame: Date treatment consent signed to date off study, approximately 109 months and 15 days and 110 months and 13 days for Arm 1 and Arm 2 respectively.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 1 - Enzalutamide Alone | Arm 2 - Enzalutamide With Prostate-Specific Antigen (PSA)-TRICOM
Number analyzed (Participants) | 29 | 28
Participants | 29 | 28

ADVERSE EVENTS:
Time Frame: Date treatment consent signed to date off study, approximately 109 months and 15 days and 110 months and 13 days for Arm 1 and Arm 2 respectively.
Arm/Group | Arm 1 - Enzalutamide Alone | Arm 2 - Enzalutamide With Prostate-Specific Antigen (PSA)-TRICOM
All-Cause Mortality (participants affected / at risk) | 9/29 | 11/28
Serious Adverse Events (participants affected / at risk) | 5/29 | 9/28
Other Adverse Events (participants affected / at risk) | 29/29 | 28/28
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm 1 - Enzalutamide Alone (N=29) | Arm 2 - Enzalutamide With Prostate-Specific Antigen (PSA)-TRICOM (N=28)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 2 (3)
Flu like symptoms (General disorders) | 1 (1) | 0 (0)
Fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 0 (0) | 1 (2)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2)
Infections and infestations - Other, acute cholecystitis (Infections and infestations) | 1 (1) | 0 (0)
Memory impairment (Nervous system disorders) | 1 (1) | 0 (0)
Nervous system disorders - Other, Myasthenia Gravis Crisis (Nervous system disorders) | 0 (0) | 1 (1)
Nervous system disorders - Other, nerve impingement was seen (Nervous system disorders) | 0 (0) | 1 (1)
Pain (General disorders) | 1 (1) | 1 (1)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Respiratory, thoracic and mediastinal disorders - Other, Pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 0 (0) | 1 (1)
Skin and subcutaneous tissue disorders - Other, squamous cell removal (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1)
Surgical and medical procedures - Other, Fusion, Laminectomy, and Tumor Resection (Surgical and medical procedures) | 0 (0) | 1 (1)
Surgical and medical procedures - Other, Surgical procedure, pacemaker implantation (Surgical and medical procedures) | 1 (1) | 0 (0)
Surgical and medical procedures - Other, percutaneous drain placement (Surgical and medical procedures) | 1 (1) | 0 (0)
Surgical and medical procedures - Other, right knee total arthroplasty (Surgical and medical procedures) | 1 (1) | 0 (0)
Thromboembolic event (Vascular disorders) | 1 (2) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0)
White blood cell decreased (Investigations) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm 1 - Enzalutamide Alone (N=29) | Arm 2 - Enzalutamide With Prostate-Specific Antigen (PSA)-TRICOM (N=28)
Alanine aminotransferase increased (Investigations) | 2 (2) | 5 (7)
Alkaline phosphatase increased (Investigations) | 2 (2) | 4 (5)
Amnesia (Nervous system disorders) | 1 (1) | 0 (0)
Anemia (Blood and lymphatic system disorders) | 12 (17) | 7 (12)
Anorexia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Anxiety (Psychiatric disorders) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Arthritis (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 2 (2) | 2 (4)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Atrial flutter (Cardiac disorders) | 1 (1) | 0 (0)
Atrioventricular block first degree (Cardiac disorders) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 3 (3) | 4 (5)
Bloating (Gastrointestinal disorders) | 1 (1) | 1 (1)
Blood bilirubin increased (Investigations) | 1 (1) | 0 (0)
Blurred vision (Eye disorders) | 0 (0) | 1 (1)
Breast pain (Reproductive system and breast disorders) | 1 (1) | 2 (3)
CD4 lymphocytes decreased (Investigations) | 0 (0) | 6 (11)
CPK increased (Investigations) | 3 (4) | 3 (3)
Cardiac disorders - Other, AV block 1st degree (Cardiac disorders) | 0 (0) | 1 (1)
Cataract (Eye disorders) | 1 (1) | 0 (0)
Chest pain - cardiac (Cardiac disorders) | 0 (0) | 1 (1)
Chest wall pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Chills (General disorders) | 0 (0) | 2 (2)
Confusion (Psychiatric disorders) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 2 (2) | 3 (3)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 2 (2)
Creatinine increased (Investigations) | 2 (4) | 2 (3)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 1 (1)
Dizziness (Nervous system disorders) | 4 (5) | 1 (1)
Dry eye (Eye disorders) | 1 (1) | 2 (2)
Dysgeusia (Nervous system disorders) | 1 (2) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Edema limbs (General disorders) | 1 (2) | 2 (2)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2)
Erectile dysfunction (Reproductive system and breast disorders) | 2 (2) | 0 (0)
Eye disorders - Other, Hx Glaucoma, pre-existing (Eye disorders) | 1 (1) | 0 (0)
Eye disorders - Other, Iritis (Eye disorders) | 1 (1) | 0 (0)
Facial nerve disorder (Nervous system disorders) | 0 (0) | 1 (2)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 2 (3)
Fatigue (General disorders) | 10 (11) | 8 (12)
Fever (General disorders) | 1 (1) | 3 (4)
Flatulence (Gastrointestinal disorders) | 0 (0) | 1 (1)
Flu like symptoms (General disorders) | 2 (2) | 7 (20)
Fracture (Injury, poisoning and procedural complications) | 2 (3) | 2 (2)
Gastritis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 1 (2)
Gastrointestinal disorders - Other, Blood in stool (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrointestinal disorders - Other, EGD procedure (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gynecomastia (Reproductive system and breast disorders) | 4 (4) | 3 (4)
Headache (Nervous system disorders) | 4 (4) | 3 (5)
Hemorrhoidal hemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Hemorrhoids (Gastrointestinal disorders) | 1 (1) | 0 (0)
Hot flashes (Vascular disorders) | 7 (7) | 4 (4)
Hypercalcemia (Metabolism and nutrition disorders) | 6 (8) | 3 (3)
Hyperglycemia (Metabolism and nutrition disorders) | 17 (40) | 16 (36)
Hyperkalemia (Metabolism and nutrition disorders) | 5 (11) | 6 (9)
Hypernatremia (Metabolism and nutrition disorders) | 5 (6) | 1 (1)
Hypertension (Vascular disorders) | 0 (0) | 3 (3)
Hyperuricemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypoalbuminemia (Metabolism and nutrition disorders) | 4 (6) | 5 (5)
Hypocalcemia (Metabolism and nutrition disorders) | 2 (2) | 1 (1)
Hypoglycemia (Metabolism and nutrition disorders) | 2 (2) | 1 (1)
Hyponatremia (Metabolism and nutrition disorders) | 1 (1) | 1 (3)
Hypophosphatemia (Metabolism and nutrition disorders) | 9 (13) | 4 (7)
Hypotension (Vascular disorders) | 0 (0) | 2 (2)
Hypothyroidism (Endocrine disorders) | 1 (1) | 0 (0)
Infections and infestations - Other, C. Difficile (Infections and infestations) | 0 (0) | 1 (1)
Infections and infestations - Other, COVID-19 infection (Infections and infestations) | 0 (0) | 1 (1)
Infections and infestations - Other, Pneumonia (Infections and infestations) | 1 (1) | 0 (0)
Infections and infestations - Other, Soft tissue infection, Cellulitis (Infections and infestations) | 1 (2) | 0 (0)
Infections and infestations - Other, thrush Nystatin helped-ongoing (Infections and infestations) | 1 (1) | 0 (0)
Injection site reaction (General disorders) | 0 (0) | 24 (124)
Injury, poisoning and procedural complications - Other, Fall (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Injury, poisoning and procedural complications - Other, Pain -injury fall (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Insomnia (Psychiatric disorders) | 2 (2) | 1 (1)
Localized edema (General disorders) | 0 (0) | 1 (1)
Lymphocyte count decreased (Investigations) | 12 (23) | 15 (32)
Memory impairment (Nervous system disorders) | 1 (2) | 2 (2)
Musculoskeletal and connective tissue disorder - Other, R. ankle sprain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Musculoskeletal and connective tissue disorder - Other, closed hip (left) reduction (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 3 (4)
Nail infection (Infections and infestations) | 1 (1) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 4 (5) | 3 (4)
Nausea (Gastrointestinal disorders) | 4 (4) | 7 (10)
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, Bladder Dysplasia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, MOHs procedure (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Nervous system disorders - Other, Myasthenia Gravis (Nervous system disorders) | 0 (0) | 1 (1)
Nervous system disorders - Other, Spinal cord compression T-6 (Nervous system disorders) | 0 (0) | 1 (1)
Neuralgia (Nervous system disorders) | 1 (2) | 1 (1)
Neutrophil count decreased (Investigations) | 5 (13) | 10 (24)
Non-cardiac chest pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Oral pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
Osteonecrosis of jaw (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (2)
Osteoporosis (Musculoskeletal and connective tissue disorders) | 3 (3) | 0 (0)
Pain (General disorders) | 9 (16) | 10 (16)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 4 (5) | 4 (5)
Paresthesia (Nervous system disorders) | 1 (1) | 1 (1)
Pelvic pain (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Peripheral motor neuropathy (Nervous system disorders) | 1 (1) | 0 (0)
Platelet count decreased (Investigations) | 3 (5) | 4 (8)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 3 (4) | 0 (0)
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
Presyncope (Nervous system disorders) | 0 (0) | 2 (3)
Proctitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Proteinuria (Renal and urinary disorders) | 1 (1) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Rash acneiform (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 3 (4) | 2 (2)
Reproductive system and breast disorders - Other, RUL infiltrates (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Respiratory, thoracic and mediastinal disorders - Other, RLL infiltrates. As noted on CT scan (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Respiratory, thoracic and mediastinal disorders - Other, URI (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Rhinitis infective (Infections and infestations) | 0 (0) | 1 (1)
Salivary gland infection (Infections and infestations) | 0 (0) | 1 (1)
Sinus bradycardia (Cardiac disorders) | 0 (0) | 1 (1)
Sinusitis (Infections and infestations) | 7 (9) | 1 (1)
Skin and subcutaneous tissue disorders - Other, Fibroma (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Skin and subcutaneous tissue disorders - Other, Fungal infection (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Skin and subcutaneous tissue disorders - Other, abrasion (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Skin and subcutaneous tissue disorders - Other, papule (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Skin infection (Infections and infestations) | 0 (0) | 1 (1)
Sneezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Surgical and medical procedures - Other, Arthroscopic (Surgical and medical procedures) | 1 (1) | 0 (0)
Surgical and medical procedures - Other, Choleycystectomy (Surgical and medical procedures) | 1 (1) | 0 (0)
Surgical and medical procedures - Other, Cystoscopy (Surgical and medical procedures) | 0 (0) | 2 (2)
Surgical and medical procedures - Other, Cytoscopy (Surgical and medical procedures) | 1 (1) | 0 (0)
Surgical and medical procedures - Other, I & D of right hand abscess (Surgical and medical procedures) | 0 (0) | 1 (1)
Surgical and medical procedures - Other, MOHs - left ear (Surgical and medical procedures) | 0 (0) | 1 (1)
Surgical and medical procedures - Other, Septoplasty (Surgical and medical procedures) | 1 (1) | 0 (0)
Surgical and medical procedures - Other, TURBT (Surgical and medical procedures) | 1 (1) | 0 (0)
Tooth infection (Infections and infestations) | 2 (2) | 1 (1)
Toothache (Gastrointestinal disorders) | 1 (1) | 2 (3)
Upper respiratory infection (Infections and infestations) | 3 (9) | 3 (3)
Urinary incontinence (Renal and urinary disorders) | 0 (0) | 1 (1)
Urinary retention (Renal and urinary disorders) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1) | 2 (2)
Urinary tract obstruction (Renal and urinary disorders) | 1 (1) | 1 (1)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1) | 4 (4)
Watering eyes (Eye disorders) | 0 (0) | 1 (1)
Weight loss (Investigations) | 1 (1) | 0 (0)
White blood cell decreased (Investigations) | 9 (13) | 13 (30)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-03-29): https://cdn.clinicaltrials.gov/large-docs/33/NCT01867333/Prot_SAP_000.pdf
  • Informed Consent Form (2020-02-07): https://cdn.clinicaltrials.gov/large-docs/33/NCT01867333/ICF_001.pdf